CLINICAL TRIAL: NCT01554774
Title: Observational Study of Comparison of Echocardiographic Markers of Right Ventricular Function and Electrocardiographic Signs of Chronic Cor Pulmonale in Elderly Patient With COPD
Brief Title: Non-invasive Assessment of Pulmonary Vascular Resistance in Elderly Patients With Chronic Obstructive Pulmonary Disease
Acronym: PVR-COPD
Status: Completed | Type: Observational
Sponsor: Hospital Viamed Valvanera, Spain (Other)
Collaborators: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Vincenzo Malafarina, MD MSc, MD MSc, Hospital Viamed Valvanera, Spain
Other Study IDs: HVVV-CBM-01
Record Dates: First submitted 2012-03-02; First posted 2012-03-15 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Hypertension; Cor Pulmonale
Keywords: COPD; PVR
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary; Pulmonary Heart Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- GOLD II: Will be included in this group the patients with COPD stage II
- GOLD III: Will be included in this group the patients with COPD stage III
- GOLD IV: Will be included in this group the patients with COPD stage VI.

SUMMARY:
Many studies have evaluated the viability of measuring the pulmonary vascular resistance (PVR) by non-invasive methods in patients with pulmonary hypertension, pulmonary thromboembolism, ischemic cardiopathy and valvular disease. The investigators have not found other studies which evaluate the PVR in elderly patients with COPD. The hypothesis is that in patients with COPD, the severity of obstruction, expressed by GOLD class, is associated with an increase of PVR.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD stage II, III or IV according to the GOLD guidelines
* signed the informed consent

Exclusion Criteria:

* ischemic cardiopathy
* severe valvular disease
* atrial fibrillation
* left bundle branch block

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of patients with a diagnosis of COPD who were treated in the consulting rooms of the department of respiratory physiopathology.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
right ventricular function and GOLD stages | cross sectional
  To compare right ventricular function, evaluated by a non-invasive method such as echocardiography, with the GOLD stages in chronic obstructive pulmonary disease (COPD) patients.

SECONDARY OUTCOMES:
Right ventricular function and FEV1. | cross sectional
  Compare right ventricular function, evaluated by a non-invasive method such as echocardiography, tricuspid annulus plane systolic excursion (TAPSE),pulmonary artery systolic pressure (PAPs) and fractional area change (FAC), with the GOLD stages in chronic obstructive pulmonary disease (COPD) patients.
ECG and echocardiography parameters of cor pulmonale | cross sectional
  The correlation between right ventricular function and the electrocardiographic parameters of cor pulmonale.
Right ventricle function and 6M-WT. | cross sectional
  Evaluate the correlation between the hemodynamic indices of right ventricle and the six minute walking test (6M-WT).

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Malafarina, MD MSC, Principal Investigator — Hospital Viamed Valvanera, Spain; Raffaele Antonelli Incalzi, MD, Study Director — Campus Bio-Medico University. S. Raffaele - Cittadella della Carità Foundation, Taranto, Italy
Locations (1):
- Campus Bio-Medico University, Roma, Italy, Italy

REFERENCES:
- [Background] Incalzi RA, Fuso L, De Rosa M, Di Napoli A, Basso S, Pagliari G, Pistelli R. Electrocardiographic signs of chronic cor pulmonale: A negative prognostic finding in chronic obstructive pulmonary disease. Circulation. 1999 Mar 30;99(12):1600-5. doi: 10.1161/01.cir.99.12.1600. PMID 10096937
- [Background] Scapellato F, Temporelli PL, Eleuteri E, Corra U, Imparato A, Giannuzzi P. Accurate noninvasive estimation of pulmonary vascular resistance by Doppler echocardiography in patients with chronic failure heart failure. J Am Coll Cardiol. 2001 Jun 1;37(7):1813-9. doi: 10.1016/s0735-1097(01)01271-2. PMID 11401116
- [Background] Abbas AE, Fortuin FD, Schiller NB, Appleton CP, Moreno CA, Lester SJ. A simple method for noninvasive estimation of pulmonary vascular resistance. J Am Coll Cardiol. 2003 Mar 19;41(6):1021-7. doi: 10.1016/s0735-1097(02)02973-x. PMID 12651052
- [Background] Bossone E, Bodini BD, Mazza A, Allegra L. Pulmonary arterial hypertension: the key role of echocardiography. Chest. 2005 May;127(5):1836-43. doi: 10.1378/chest.127.5.1836. PMID 15888866
- [Background] Milan A, Magnino C, Veglio F. Echocardiographic indexes for the non-invasive evaluation of pulmonary hemodynamics. J Am Soc Echocardiogr. 2010 Mar;23(3):225-39; quiz 332-4. doi: 10.1016/j.echo.2010.01.003. PMID 20206827
- [Background] Haddad F, Zamanian R, Beraud AS, Schnittger I, Feinstein J, Peterson T, Yang P, Doyle R, Rosenthal D. A novel non-invasive method of estimating pulmonary vascular resistance in patients with pulmonary arterial hypertension. J Am Soc Echocardiogr. 2009 May;22(5):523-9. doi: 10.1016/j.echo.2009.01.021. PMID 19307098
- [Background] Kim SH, Yi MZ, Kim DH, Song JM, Kang DH, Lee SD, Song JK. Prognostic value of echocardiographic estimation of pulmonary vascular resistance in patients with acute pulmonary thromboembolism. J Am Soc Echocardiogr. 2011 Jun;24(6):693-8. doi: 10.1016/j.echo.2011.02.002. Epub 2011 Mar 24. PMID 21439783
- [Background] Farzaneh-Far R, Na B, Whooley MA, Schiller NB. Usefulness of noninvasive estimate of pulmonary vascular resistance to predict mortality, heart failure, and adverse cardiovascular events in Patients With stable coronary artery disease (from the Heart and Soul Study). Am J Cardiol. 2008 Mar 15;101(6):762-6. doi: 10.1016/j.amjcard.2007.11.010. Epub 2008 Feb 21. PMID 18328836
- [Background] Choi EY, Shim J, Kim SA, Shim CY, Yoon SJ, Kang SM, Choi D, Ha JW, Rim SJ, Jang Y, Chung N. Value of echo-Doppler derived pulmonary vascular resistance, net-atrioventricular compliance and tricuspid annular velocity in determining exercise capacity in patients with mitral stenosis. Circ J. 2007 Nov;71(11):1721-7. doi: 10.1253/circj.71.1721. PMID 17965491
- [Background] Arcasoy SM, Christie JD, Ferrari VA, Sutton MS, Zisman DA, Blumenthal NP, Pochettino A, Kotloff RM. Echocardiographic assessment of pulmonary hypertension in patients with advanced lung disease. Am J Respir Crit Care Med. 2003 Mar 1;167(5):735-40. doi: 10.1164/rccm.200210-1130OC. Epub 2002 Dec 12. PMID 12480614
- [Background] Barbera JA, Peinado VI, Santos S. Pulmonary hypertension in chronic obstructive pulmonary disease. Eur Respir J. 2003 May;21(5):892-905. doi: 10.1183/09031936.03.00115402. PMID 12765440
- [Background] Burgess MI, Ray S, Mogulkoc N, Egan J, Incalzi RA, Fuso L, Marino De Rosa, Di Napoli A, Basso S, Pagliari G, Pistelli R. Doppler echocardiographic index of global right ventricular function. Circulation. 2000 Mar 28;101(12):E117. doi: 10.1161/01.cir.101.12.e117. No abstract available. PMID 10736299